CLINICAL TRIAL: NCT01536912
Title: Behavioral Economic Analysis of Medical Marijuana Use in HIV+ Patients: Probability Survey
Brief Title: Medical Marijuana Use in HIV+ Patients: Probability Survey
Acronym: MMS
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor, Wayne State University
Other Study IDs: MMS-1; R01DA032678 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: HIV Positive
Keywords: HIV positive
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
More scientific information is needed about medical marijuana use among HIV positive patients. There is conflicting information about the use of marijuana, use of medical marijuana, and the associations between them and health status/health risk behaviors/health care utilization. In addition, it is not clear whether patients who participate in prospective clinical studies differ from participants who do not participate; if there are differences between those two groups, then this would limit generalizability of knowledge about these issues.

The goal of this project is to describe the use of marijuana among HIV positive patients and its association with health status/health risk behaviors/health care utilization.

DETAILED DESCRIPTION:
Participants will answer questions about marijuana, medical marijuana, and other drug use. We will also ask about health and steps participants take to keep healthy. The study will take up to one hour to complete.

Participants will also be asked to sign a release of information form. This form would allow us to look at medical records at the HIV clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the HIV clinic
* HIV positive

Exclusion Criteria:

* Lack of english

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University (HIV clinic, Tolan Park Medical Building), Detroit, Michigan, United States